CLINICAL TRIAL: NCT00536783
Title: Schizophrenia Sensory Gating Deficit With Quetiapine
Status: Completed | Type: Observational
Sponsor: New Mexico VA Healthcare System (U.S. Federal Agency)
Collaborators: AstraZeneca (Industry)
Other Study IDs: 0072; . IRUSQUET0332
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2007-12-31 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia
Keywords: Psychiatry; Antipsychotic; Psychopharmacology; Clinical Trial; Open Label; Schizophrenia; Sensory Gating; Attention; Memory
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The purpose of this study is the use of magnetoencephalography or MEG (a machine that measures magnetic activity in your brain) and electroencephalography or EEG (a technique that measures electrical activity in your brain) to study how sounds are processed in individuals with schizophrenia after three months of taking the antipsychotic medication quetiapine.

DETAILED DESCRIPTION:
.Problems with attention and perception are core features of schizophrenia and are hypothesized to result from defects in the filtering or gating of sensory input. Examination of this requires neuoimaging techniques with high temporal resolution. High-density EEG and MEG in combination with structural magnetic resonance imaging (sMRI) are used to map sensory gating. In a number of recent studies patient treated with novel antipsychotics have been shown to have P50 gating ratios resembling those of normal controls rather than that of schizophrenia subjects treatment with conventional antipsychotics. To date, there is no literature on the effects of quetiapine on sensory gating. Subjects who meet all inclusion criteria and have been on a stable dose of quetiapine for three months will receive a clinical interview, an MRI, MEG, and neuropsychological testing to determine if patients with schizophrenia who are treated with quetiapine will demonstrate a sensory gating ratio similar to normal controls, indicating no deficit in sensory gating.

ELIGIBILITY:
Inclusion Criteria:

Patient Population

* Diagnosis of Schizophrenia as determine by the Structured Clinical Interview for DSM-IV
* No comorbid diagnosis of PTSD
* responders to quetiapine, determined by continuous treatment at the same dose of quetiapine and absence of psychiatric hospitalization for at least 3 months
* No history of drug dependency in their lifetime
* No history of alcohol or other substance abuse in the 6 months prior to entry into the study
* No history of head injury with loss of consciousness for more than 5 minutes
* No history of seizure disorder
* No mood stabilizing agents
* Between 18-65 and
* Able to sign informed consent

Normal Controls

* Matched in age and gender to patient population
* No history of psychiatric dysfunction or alcohol or other substance dependence in their lifetime as determine by the SCID
* No history of alcohol or other substance abuse in the previous 6 months
* No family history of psychotic disorder in first degree relatives as assessed by the FH-RDC diagnostic interview
* No history of head injury with loss of consciousness for more than 5 minutes
* No history of seizure disorder
* Between 18-65
* Able to sign informed consent

Exclusion Criteria:

Subjects will be excluded from participating in this study if they:

* Require treatment with a mood stabilizer
* Have had an inpatient hospitalization in the past 3 months
* Have a history of a neurological disorder
* Have any other axis I diagnosis besides schizophrenia

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-04; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Canive, MD, Principal Investigator — New Mexico VA Heathcare System / BRINM
Locations (1):
- New Mexico VA Healthcare System, Albuquerque, New Mexico, United States

REFERENCES:
- See also: The website for the Biomedical Research Institute of New Mexico which helps administers the funds for this project. — http://www.brinm.org